## STATISTICAL ANALYSIS PLAN COVER PAGE

Study Title:

Effects of a Physical Activity Program for Children with Autism on Psychomotor and Psychosocial Characteristics

Principal Investigator: Ebru AYAZ

Independent Researcher / Kocaeli – Turkey

E-mail: ebrukaracar41@hotmail.com

Orcid: https://orcid.org/0009-0006-7186-9178

Second Author: Dilara Fatoş ÖZER

Istanbul Bilgi University / Faculty of Health Sciences - Department of Child Development /

Istanbul – Turkey

E-mail: dilara.ozer@bilgi.edu.tr

Orcid: https://orcid.org/0000-0001-5753-3332

Third Author: Gülsüm HATİPOĞLU ÖZCAN

Istanbul University-Cerrahpaşa / Faculty of Sport Sciences / Istanbul – Turkey

E-mail: gulsumhatipoglu@hotmail.com

Orcid: https://orcid.org/0000-0003-1059-8424

NCT Number: Not Yet Appointed

Document Type: Statistical Analysis Plan

Document Date: 10/04/2022

## STATISTICAL ANALYSIS PLAN

SPSS (Statistical Package for the Social Sciences) 25.0 will be used for statistical analysis of the data. In addition to descriptive statistical methods (Mean, Standard Deviation, Median, Frequency, Ratio, Minimum, Maximum), the Kolmogorov-Smirnov test will be performed to determine whether the data are normally distributed. Data analysis using the Mann-Whitney U test and Wilcoxon signed-rank test aimed to determine statistically significant differences between the GARS-2 TV, BOT-2, SSRS-PF, Eurofit, and PedsQL test scores obtained before and after the 10-week PAP. The Mann-Whitney U test will be used for two-group comparisons of parameters that do not show a normal distribution, and the Wilcoxon signed-rank test will be used to examine changes between pretest and posttest measurements. Effect size values (Cohen's d and r) will be calculated to assess the magnitude of the effect of PAP on the variables. Significance will be assessed at p<0.05.

Thematic analysis method will be used for the focus group interview, which is one of the qualitative research methods.